CLINICAL TRIAL: NCT06808646
Title: A Phase 1, Single-center, Open-label, Non-randomized, Fixed-sequence, Drug-drug Interaction Study to Assess the Effect of Repeated Doses of Intravenous Ceftobiprole on the Pharmacokinetics of Oral Pitavastatin (OATP1B Substrate) and on Plasma Levels of Coproporphyrin I (OATP1B Biomarker) in Healthy Subjects
Brief Title: A Study to Assess the Effect of Ceftobiprole on the PK of Pitavastatin and on Plasma Levels of Coproporphyrin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: BPR-CP-101
Record Dates: First submitted 2025-01-09; First posted 2025-02-05 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Drug-drug Interaction Study
Keywords: Ceftobiprole; Pitavastatin; OATP1B; Coproporphyrin; DDI
MeSH Terms: interventions — pitavastatin; ceftobiprole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Period 1; pitavastatin single dose, Period 2; pitavastatin single dose combined with ceftobiprole (Experimental): Period 1 On Day 1, a single oral dose of pitavastatin will be administered
  Period 2 From Day 4 to Day 7, ceftobiprole (as the prodrug ceftobiprole medocaril sodium) will be administered intravenously (IV) every 8 hours (q8h) for four days. On Day 6, a single oral dose of pitavastatin will be co-administered with ceftobiprole
  Interventions: Drug: pitavastatin; Drug: pitavastatin single dose combined with ceftobiprole

INTERVENTIONS:
Drug: pitavastatin — Single oral administration
Drug: pitavastatin single dose combined with ceftobiprole — Single oral pitavastatin co-administered with IV ceftobiprole

SUMMARY:
The goal of this clinical study is to determine the effect of the test drug ceftobiprole (a drug approved for the treatment of bacterial infections) on the elimination of pitavastatin (a drug approved for the treatment of increased levels of cholesterol in blood) from the body. This interaction will be investigated by pharmacokinetic (PK) assessments.

The PK of pitavastatin will be assessed when administered alone and when administered together with ceftobiprole in a study design including two treatment periods.

The clinical study will also investigate the safety of ceftobiprole and how well ceftobiprole is tolerated by healthy subjects when it is administered in combination with pitavastatin. In addition, the effect of ceftobiprole on a specific marker, called coproporphyrin I, will be assessed in the blood.

The duration of the study will be a maximum of 38 days.

ELIGIBILITY:
Main Inclusion Criteria:

* Body mass index: 18.0 to 30.0 kg/m2, inclusive
* Good physical and mental health
* Normal renal function (creatinine clearance ≥ 90 mL/min as determined by the Cockcroft-Gault equation)
* Female participants of childbearing potential must not be pregnant or lactating and must must agree to use adequate contraception
* Male subjects, if not surgically sterilized, must agree to use adequate contraception
* All prescribed medication must have been stopped at least 30 days prior to admission to the clinical research center (an exception is made for hormonal contraceptives)
* All over-the-counter medication, vitamin preparations and other food supplements, or herbal medications (e.g., St. John's wort) must have been stopped at least 14 days prior to admission to the clinical research center
* Ability and willingness to abstain from alcohol from 48 hours (2 days) prior to Screening and admission to the clinical research center
* Ability and willingness to abstain from methylxanthine-containing beverages or food from 48 hours (2 days) prior to admission to the clinical research center

Main Exclusion Criteria:

* History of relevant drug and/or food allergies, particularly to antibiotics.
* Subject received a known potent inhibitor of OATP1B activity within 30 days prior to admission
* Subject received a potential inducer of OATP1B activity within 30 days prior to admission
* Subject has a history of seizures
* Subject has a history of frequent diarrhea
* Smoking more than 5 cigarettes, 1 cigar, or 1 pipe daily; the use of tobacco products in the 48 hours (2 days) prior to admission
* History of alcohol abuse or drug addiction within 12 months prior to Screening.
* Average intake of more than 24 units of alcohol per week
* Positive drug and/or alcohol screen
* Donation or loss of more than 450 mL of blood within 60 days prior to the first pitavastatin administration on Day 1 of the current study. Donation or loss of more than 1.5 liters of blood (for male subjects)/more than 1.0 liters of blood (for female subjects) in the 10 months prior to the first pitavastatin administration on Day 1 of the current study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) after a single oral dose of pitavastatin administered without and with intravenous (IV) ceftobiprole | Up to Day 8
Area under the plasma concentration-time curve up to time (AUC0-t) after a single oral dose of pitavastatin administered without and with IV ceftobiprole | Up to Day 8
Area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf) after a single oral dose of pitavastatin administered without and with IV ceftobiprole | Up to Day 8

SECONDARY OUTCOMES:
Cmax of coproporphyrin I (CP-I) after IV ceftobiprole administration | Up to Day 8
Area under the plasma level-time curve up to time 25.5 hours (AUEC0-25.5h) of CP-I after IV ceftobiprole administration | Up to Day 8
Cmax of IV ceftobiprole without and with oral administration of pitavastatin | Up to Day 8
Area under the plasma concentration-time curve up to 8 hours (AUC0-8h) after IV ceftobiprole without and with oral administration of pitavastatin | Up to Day 8
Cmax of the pitavastatin metabolite pitavastatin lactone after a single oral dose of pitavastatin, administered without and with IV ceftobiprole | Up to Day 8
AUC0-t of the pitavastatin metabolite pitavastatin lactone after a single oral dose of pitavastatin, administered without and with IV ceftobiprole | Up to Day 8
AUC0-inf of the pitavastatin metabolite pitavastatin lactone after a single oral dose of pitavastatin, administered without and with IV ceftobiprole | Up to Day 8
Number of participants reporting Treatment-emergent adverse events (TEAEs) after administration of ceftobiprole without and with a single oral dose of pitavastatin | Up to Day 17
Number of participants with clinically significant change from baseline in laboratory parameters after administration of ceftobiprole without and with a single oral dose of pitavastatin | Up to Day 17
Number of participants with clinically significant change from baseline in vital signs after administration of ceftobiprole without and with a single oral dose of pitavastatin | Up to Day 17
Number of participants with clinically significant change from baseline in 12-lead electrocardiogram (ECG) parameters after administration of ceftobiprole without and with a single oral dose of pitavastatin | Up to Day 17

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kaindl, MD, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (1):
- ICON Early Clinical & Bioanalytical Solutions, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-12-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT06808646/ICF_000.pdf